CLINICAL TRIAL: NCT00537602
Title: Single Center, Double-blind, Randomized, Placebo-controlled, 2-period/2-treatment Crossover Study Investigating the Effect of Miglustat on the Nasal Potential Difference in Patients With Cystic Fibrosis Homozygous for the ΔF508 Mutation
Brief Title: Miglustat / OGT 918 in the Treatment of Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Methodology applied did not meet all criteria required per guidelines
Sponsor: Actelion (Industry)
Responsible Party: Paul van Giersbergen , PhD, Actelion
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-056-201
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; miglustat; Zavesca; Actelion; nasal potential difference; transmembrane conductance regulator (CFTR)
MeSH Terms: conditions — Cystic Fibrosis | interventions — miglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Oral miglustat capsules 200 mg t.i.d. for 1 week and a single 200 mg dose on day 8
  Interventions: Drug: miglustat
- B (Placebo Comparator): Oral placebo capsules matching in appearance miglustat capsules given t.i.d. for 1 week and a single dose on day 8
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: miglustat
  Other Names: Zavesca; OGT 918; 1.5- (Butylimino) -1.5- Dideoxy-D-Glucitol
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
Cystic fibrosis is a genetic disease caused by mutation of the cystic fibrosis transmembrane conductance regulator (CFTR). The purpose of the study is to investigate the effects of miglustat on CFTR function in cystic fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 years and older
* Male or female
* Non-pregnant women who are to remain non-pregnant for 3 months after the end of the study: only women who are surgically sterile, who are in the menopause (no menstruation for at least one year) or those of childbearing potential who are using a reliable method of contraception. Reliable methods of contraception for female patients include the following:

  * Barrier type devices (e.g., female condom, diaphragm and contraceptive sponge) used ONLY in combination with a spermicide
  * Intrauterine devices
  * Oral contraceptive agent
  * Depo-Provera™ (medroxyprogesterone acetate)
  * Levonorgestrel implants Abstention, the rhythm method or contraception by the partner alone are NOT reliable methods of contraception.

For children, a reliable method of contraception must be considered, if appropriate.

* Accepting for the duration of the study and for 3 months thereafter to use a condom and not to procreate a child (males only)
* Cystic fibrosis patients homozygous for the ΔF508 mutation as confirmed by genetic test
* Signed informed consent prior to any study-mandated procedure

Exclusion Criteria:

* Any condition prohibiting the correct measurement of the NPD such as upper respiratory tract infection
* Acute upper respiratory tract or pulmonary exacerbation requiring antibiotic intervention within 2 weeks of screening
* Severe renal impairment (creatinine clearance < 30 ml/min as per Cockroft and Gault)
* Female patients who will not undergo a pregnancy test prior to enrollment in the study
* History of significant lactose intolerance
* History of neuropathy
* History of cataracts or known increased risk of cataract formation
* Presence of clinically significant diarrhea (>3 liquid stolls per days for >7 days) without definable cause within 1 month prior to screening
* Any known factor of disease that might interfere with treatment compliance, study conduct or interruption of the results such as drug or alcohol dependence or psychiatric disease
* FEVI <25% of predicted normal
* Oxygen saturation at rest <88%
* Active or passive smoking as measured using the Smokelyzer®
* Hypersensitivity to miglustat or any excipients
* Planned treatment or treatment with another investigational drug or therapy (e.g., gene therapy) within 1 month prior to randomization

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in nasal potential difference (NPD) in response to isoproterenol in chloride-free buffer in the presence of amiloride | Baseline (pre-dose on day 1) to end-of-treatment (day 8)

SECONDARY OUTCOMES:
Change in baseline NPD response | Baseline to end-of-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul van Giersbergen, PhD, Study Director — Actelion; Christian Domingo-Ribas, MD, Principal Investigator — Corporacio Parc Tauli
Locations (1):
- Corporacio Parc Tauli / Parc Tauli Hospital, Barcelona, Spain